CLINICAL TRIAL: NCT03668886
Title: A Multimodal Exercise Program in Musculoskeletal System of the Community Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2001800707B0
Record Dates: First submitted 2018-08-29; First posted 2018-09-13 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2018-08

CONDITIONS: Elderly Exercise

STUDY DESIGN:
Intervention Model Description: intervention group: receive multimodal exercise program for half year control group: participate community activity
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multimodal exercise program (Experimental): Elderly in this group will receive multimodal exercise program. The duration of exercise is 60 minutes and frequency is 2 times/week.
  Interventions: Other: multimodal exercise program
- Control group (No Intervention): Elderly in this group will continue to attend community activity as usual. The activity includes active activity is 60 minutes and frequency is 2 times/week.

INTERVENTIONS:
Other: multimodal exercise program — warm-up, strengthening exercise, aerobic exercise, cool-down
  Arms: multimodal exercise program

SUMMARY:
The number of elderly has been increasing in recent decades. Current studies focused on the risk factors of poor physical performance, poor daily activity performance, and even disability in the elderly. We planned to evaluate the physical performance of elderly dwelling in the community and designed a multimodal exercise program which can improve physical performance, prevent disability and promote quality of life.

ELIGIBILITY:
Inclusion Criteria:

* >= 65 year old

Exclusion Criteria:

* cognitive impairment and poor understanding for orders
* the elderly has medical problems that the elderly can't perform exercise

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Gait speed | change between two time points (baseline, 3 months later)
  measure gait speed as usual
Gait speed | change between two time points (baseline, 6 months later)
  measure gait speed as usual

SECONDARY OUTCOMES:
Muscle mass | change between two time points (baseline, 6 months later)
  Measure by body composition study
Level (mild, moderate, maximal) of daily activity | change between two time points (baseline, 3 months later)
  Use pedometer
Level (mild, moderate, maximal) of daily activity | change between two time points (baseline, 6 months later)
  Use pedometer
Zipper test | change between two time points (baseline, 3 months later)
  use for evaluation of flexibility
Zipper test | change between two time points (baseline, 6 months later)
  use for evaluation of flexibility
Sit and reach test | change between two time points (baseline, 3 months later)
  use for evaluation of flexibility
Sit and reach test | change between two time points (baseline, 6 months later)
  use for evaluation of flexibility
Biceps strength | change between two time points (baseline, 3 months later)
  Times of biceps curls within 30 seconds
Biceps strength | change between two time points (baseline, 6 months later)
  Times of biceps curls within 30 seconds
Strength of lower limbs | change between two time points (baseline, 3 months later)
  Times of sit and stand test within 30 seconds
Strength of lower limbs | change between two time points (baseline, 6 months later)
  Times of sit and stand test within 30 seconds
One leg stand test | change between two time points (baseline, 3 months later)
  measure the duration when standing on one leg
One leg stand test | change between two time points (baseline, 6 months later)
  measure the duration when standing on one leg
Timed up and go test | change between two time points (baseline, 3 months later)
  measure the time spent for standing up, walking for 3 meter, turning around, going back and sitting down
Timed up and go test | change between two time points (baseline, 6 months later)
  measure the time spent for standing up, walking for 3 meter, turning around, going back and sitting down
Endurance | change between two time points (baseline, 3 months later)
  6 minutes walking test
Endurance | change between two time points (baseline, 6 months later)
  6 minutes walking test
Range of motion of knee | change between two time points (baseline, 3 months later)
  measure by goniometer
Range of motion of knee | change between two time points (baseline, 6 months later)
  measure by goniometer
Pain, stiffness, physical function of knee | change between two time points (baseline, 3 months later)
  WOMAC (Western Ontario and McMaster Universities Arthritis Index) questionnaire is used for evaluation of pain, stiffness, physical function of patients with knee osteoarthritis. It includes 5 questions for pain, 2 questions for stiffness and 17 questions for physical function. The score of every question is from 0 to 4. The larger the number, the discomfort becomes more servere. We use the difference of change between two time points (baseline, 3 months later) to measure the benefit of the exercise.
Pain, stiffness, physical function of knee | change between two time points (baseline, 6 months later)
  WOMAC (Western Ontario and McMaster Universities Arthritis Index) questionnaire is used for evaluation of pain, stiffness, physical function of patients with knee osteoarthritis. It includes 5 questions for pain, 2 questions for stiffness and 17 questions for physical function. The score of every question is from 0 to 4. The larger the number, the discomfort becomes more servere. We use the difference of change between two time points (baseline, 6 months later) to measure the benefit of the exercise.
Grip strength | change between two time (baseline, 3 months later)
  measure grip strength by Camry EH101
Grip strength | change between two time (baseline, 6 months later)
  measure grip strength by Camry EH101

CONTACTS AND LOCATIONS:
Overall Officials: Shui Tseng, Study Chair — Chang Gung Medical Foundation Institutional Review Board
Locations (1):
- Yu Hsuan Tseng, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No